CLINICAL TRIAL: NCT01817491
Title: Low Fat Vegan Diet or American Heart Association Diet, Impact on Biomarkers of Inflammation, Oxidative Stress and Cardiovascular Risk in Obese 9-18 y.o. With Elevated Cholesterol: A Four Week Randomized Trial
Brief Title: Low Fat Vegan or American Heart Association Diets & Cardiovascular Risk in Obese 9-18 y.o. With Elevated Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, michael macknin, Professor of Pediatrics Cleveland Clinic Lerner College of Medicine of Case Western Reserve, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1298
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Disease; Hypercholesterolemia; Obesity; Fatty Liver
Keywords: Vegan Diet; Hypercholesterolemia; American Heart Association Diet; Cardiovascular Risk; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Obesity; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced Fat Vegan Diet (Active Comparator): Plant based diet with as few added oils and fats as possible.
  Interventions: Other: Reduced Fat Vegan Diet
- American Heart Association Diet (Active Comparator): Diet emphasizing fruits, vegetables and whole grains but also low fat dairy, low fat meat and fish.
  Interventions: Other: American Heart Association Diet

INTERVENTIONS:
Other: American Heart Association Diet
  Arms: American Heart Association Diet
Other: Reduced Fat Vegan Diet
  Arms: Reduced Fat Vegan Diet

SUMMARY:
The purpose of this study is to investigate the short-term effects of a reduced fat plant-based diet on biomarkers of inflammation, oxidative stress and cardiovascular risk. This plant-based diet consists of whole grains, fruits and vegetables and little amounts of nuts and seeds, with no limitations on the amount of food intake. Animal products are not allowed. The results of the plant-based diet will be compared with the diet recommended by American Heart Association. This diet also emphasizes fruits and vegetables, but allows healthy fats, low-fat meats, fish and low-fat dairy in moderation. The results of the study might be useful in understanding whether or not plant-based diets are protective against cardiovascular disease.

DETAILED DESCRIPTION:
Scientific Question: In obese, hypercholesterolemic (>169 mg/dl) 9-18 year olds and one of their parents are biomarkers of inflammation, oxidative stress and cardiovascular risk significantly reduced after a randomized 4 week trial of a reduced fat, vegan diet, or the American Heart Association (AHA) diet (which also encourages fruits, vegetables and whole grains, but permits low fat meat and dairy, and fish)? Rationale: "Cardiovascular disease remains the leading cause of death in North Americans, but manifest disease in childhood and adolescence is rare. By contrast, risk factors and risk behaviors that accelerate the development of atherosclerosis begin in childhood, and there is increasing evidence that risk reduction delays progression toward clinical disease". Myeloperoxidase is an early biomarker of inflammation, oxidative stress and cardiovascular risk in prepubertal obese children and is over expressed in children with hypercholesterolemia. Trimethylamine N-oxide, global arginine bioavailability ratio, arginine methylation index, paraoxonase 1 gene, and F2-isoprostane are all also associated with future major adverse cardiovascular events. Studies have suggested that a low-fat, vegan diet is effective in promoting weight loss, lowering body mass index, improving lipoprotein profiles, insulin sensitivity and in preventing cardiovascular disease in overweight individuals. Vegetarian diets have been shown to not only prevent but also to reverse heart disease in adults. Dietary habits (e.g. vegan/vegetarian versus omnivore/carnivore) are associated with significant alterations in intestinal microbiota composition and function. The diet-microbe interaction may play a significant role in the cardiovascular protective effects of a vegan/vegetarian diet. One small report of 15 adults on a reduced fat, vegan "Engine 2 Diet" for four weeks reported decreases in mean total cholesterol from 197 mg/dl to 135 mg/dl and mean LDL cholesterol falling from 124 mg/dl to 74 mg/dl.

Innovation: This is the first randomized trial comparing a low fat vegan diet to the standard AHA diet. If one diet proves superior in this brief pilot study, future larger long term studies will be needed to clearly define the health implications of our results.

Methods: Obese hypercholesterolemic children ages 9-18 will be identified by reviewing medical records and recruited initially by letters. Child, parent/guardian pairs will be randomly assigned to either the reduced fat vegan diet or the AHA diet.

During the 4-week study, participants will be asked to attend a group teaching and cooking session once a week on Saturday to learn about their assigned diets. The participants will also be requested to record their diet history on 2 weekdays and 1 weekend day before and again during the 4 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 9-18
* BMI > 95th percentile
* Hypercholesterolemia (>169 mg/dl)

Exclusion Criteria:

* Pregnant women
* Patients already on vegetarian diets

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Macknin, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Expert Panel on Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents; National Heart, Lung, and Blood Institute. Expert panel on integrated guidelines for cardiovascular health and risk reduction in children and adolescents: summary report. Pediatrics. 2011 Dec;128 Suppl 5(Suppl 5):S213-56. doi: 10.1542/peds.2009-2107C. Epub 2011 Nov 14. No abstract available. PMID 22084329
- [Background] Olza J, Aguilera CM, Gil-Campos M, Leis R, Bueno G, Martinez-Jimenez MD, Valle M, Canete R, Tojo R, Moreno LA, Gil A. Myeloperoxidase is an early biomarker of inflammation and cardiovascular risk in prepubertal obese children. Diabetes Care. 2012 Nov;35(11):2373-6. doi: 10.2337/dc12-0614. Epub 2012 Aug 21. PMID 22912422
- [Background] Pignatelli P, Loffredo L, Martino F, Catasca E, Carnevale R, Zanoni C, Del Ben M, Antonini R, Basili S, Violi F. Myeloperoxidase overexpression in children with hypercholesterolemia. Atherosclerosis. 2009 Jul;205(1):239-43. doi: 10.1016/j.atherosclerosis.2008.10.025. Epub 2008 Nov 6. PMID 19081093
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Tang WH, Wang Z, Cho L, Brennan DM, Hazen SL. Diminished global arginine bioavailability and increased arginine catabolism as metabolic profile of increased cardiovascular risk. J Am Coll Cardiol. 2009 Jun 2;53(22):2061-7. doi: 10.1016/j.jacc.2009.02.036. PMID 19477356
- [Background] Wang Z, Tang WH, Cho L, Brennan DM, Hazen SL. Targeted metabolomic evaluation of arginine methylation and cardiovascular risks: potential mechanisms beyond nitric oxide synthase inhibition. Arterioscler Thromb Vasc Biol. 2009 Sep;29(9):1383-91. doi: 10.1161/ATVBAHA.109.185645. Epub 2009 Jun 18. PMID 19542023
- [Background] Bhattacharyya T, Nicholls SJ, Topol EJ, Zhang R, Yang X, Schmitt D, Fu X, Shao M, Brennan DM, Ellis SG, Brennan ML, Allayee H, Lusis AJ, Hazen SL. Relationship of paraoxonase 1 (PON1) gene polymorphisms and functional activity with systemic oxidative stress and cardiovascular risk. JAMA. 2008 Mar 19;299(11):1265-76. doi: 10.1001/jama.299.11.1265. PMID 18349088
- [Background] Zhang ZJ. Systematic review on the association between F2-isoprostanes and cardiovascular disease. Ann Clin Biochem. 2013 Mar;50(Pt 2):108-14. doi: 10.1258/acb.2012.011263. Epub 2012 Sep 27. PMID 23019600
- [Background] Fung TT, Rimm EB, Spiegelman D, Rifai N, Tofler GH, Willett WC, Hu FB. Association between dietary patterns and plasma biomarkers of obesity and cardiovascular disease risk. Am J Clin Nutr. 2001 Jan;73(1):61-7. doi: 10.1093/ajcn/73.1.61. PMID 11124751
- [Background] Newby PK. Plant foods and plant-based diets: protective against childhood obesity? Am J Clin Nutr. 2009 May;89(5):1572S-1587S. doi: 10.3945/ajcn.2009.26736G. Epub 2009 Mar 25. PMID 19321559
- [Background] Turner-McGrievy GM, Barnard ND, Scialli AR. A two-year randomized weight loss trial comparing a vegan diet to a more moderate low-fat diet. Obesity (Silver Spring). 2007 Sep;15(9):2276-81. doi: 10.1038/oby.2007.270. PMID 17890496
- [Background] Hu FB. Plant-based foods and prevention of cardiovascular disease: an overview. Am J Clin Nutr. 2003 Sep;78(3 Suppl):544S-551S. doi: 10.1093/ajcn/78.3.544S. PMID 12936948
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Ley RE, Hamady M, Lozupone C, Turnbaugh PJ, Ramey RR, Bircher JS, Schlegel ML, Tucker TA, Schrenzel MD, Knight R, Gordon JI. Evolution of mammals and their gut microbes. Science. 2008 Jun 20;320(5883):1647-51. doi: 10.1126/science.1155725. Epub 2008 May 22. PMID 18497261
- [Background] Muegge BD, Kuczynski J, Knights D, Clemente JC, Gonzalez A, Fontana L, Henrissat B, Knight R, Gordon JI. Diet drives convergence in gut microbiome functions across mammalian phylogeny and within humans. Science. 2011 May 20;332(6032):970-4. doi: 10.1126/science.1198719. PMID 21596990
- [Background] Zimmer J, Lange B, Frick JS, Sauer H, Zimmermann K, Schwiertz A, Rusch K, Klosterhalfen S, Enck P. A vegan or vegetarian diet substantially alters the human colonic faecal microbiota. Eur J Clin Nutr. 2012 Jan;66(1):53-60. doi: 10.1038/ejcn.2011.141. Epub 2011 Aug 3. PMID 21811294
- [Background] Fraser GE. Vegetarian diets: what do we know of their effects on common chronic diseases? Am J Clin Nutr. 2009 May;89(5):1607S-1612S. doi: 10.3945/ajcn.2009.26736K. Epub 2009 Mar 25. PMID 19321569
- [Background] Rak K, Rader DJ. Cardiovascular disease: the diet-microbe morbid union. Nature. 2011 Apr 7;472(7341):40-1. doi: 10.1038/472040a. No abstract available. PMID 21475185
- [Background] Esselstyn R. The Engine 2 Diet How It All Began. In Esselstyn R "The Engine 2 Diet". New York, Boston: Wellness Central Hachette Book Group, 2009:15-30
- [Derived] Macknin M, Kong T, Weier A, Worley S, Tang AS, Alkhouri N, Golubic M. Plant-based, no-added-fat or American Heart Association diets: impact on cardiovascular risk in obese children with hypercholesterolemia and their parents. J Pediatr. 2015 Apr;166(4):953-9.e1-3. doi: 10.1016/j.jpeds.2014.12.058. Epub 2015 Feb 12. PMID 25684089

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced Fat Vegan Diet: Plant based diet with as few added oils and fats as possible.
  Reduced Fat Vegan Diet
- American Heart Association Diet: Diet emphasizing fruits, vegetables and whole grains but also low fat dairy, low fat meat and fish.
  American Heart Association Diet
Period: Overall Study
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Started | 32 | 28
Completed | 28 | 28
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 14 | 30
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years]
  Adolescents | 15 [9.0 to 18.0] | 15 [9.0 to 18.0] | 15 [9.0 to 18.0]
  Parents | 46.5 [37.0 to 61.0] | 46.0 [35.0 to 51.0] | 46.25 [35.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index BMI Percentile
Time Frame: baseline, 4 weeks
Population: Children only
Measure: Mean (Standard Deviation); unit: BMI percentile
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
BMI percentile
  Children | -1.12 (1.69) | -0.08 (0.42)
  Parents | -1.29 (1.14) | -0.73 (0.92)

2. Primary Outcome: Children Change in BMI Z Score
Description: Body mass index z-scores, also called BMI standard deviation (s.d.) scores, are measures of relative weight adjusted for child age and sex. Given a child's age, sex, BMI, and an appropriate reference standard, a BMI z-score (or its equivalent BMI-for-age percentile) can be determined. Negative BMI z-scores indicate a BMI that is lower than the population mean, while positive BMI scores indicate a value that is higher than the population mean. A decrease in the BMI z-score over time indicate a lowering of the BMI. Z-scores of 1.03 and 1.64 correspond to the 85th and 95th percentiles of BMI-for-age, which are the definitions of overweight and obesity in children.
Time Frame: baseline, 4 weeks
Population: Children only
Measure: Mean (Standard Deviation); unit: Z Score
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 14 | 14
Z Score | -0.14 (0.16) | -0.03 (0.07)

3. Primary Outcome: Change in Blood Pressure (BP)
Time Frame: baseline, 4 weeks
Population: Children and parents
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
mm Hg
  Children Systolic BP: number analyzed (Participants) | 14 | 14
  Children Systolic BP | -6.43 (8.86) | -5.14 (17.64)
  Parents Systolic BP: number analyzed (Participants) | 14 | 14
  Parents Systolic BP | -7.96 (12.28) | -3.14 (14.42)
  Children Diastolic BP: number analyzed (Participants) | 14 | 14
  Children Diastolic BP | -2.61 (10.25) | -4.36 (14.67)
  Parent Diastolic BP: number analyzed (Participants) | 14 | 14
  Parent Diastolic BP | -3.46 (11.06) | -6.64 (12.19)

4. Primary Outcome: Change in Weight
Time Frame: baseline, 4 weeks
Population: Children and parents
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
kg
  Children: number analyzed (Participants) | 14 | 14
  Children | -3.05 (3.27) | -1.55 (1.83)
  Parents: number analyzed (Participants) | 14 | 14
  Parents | -3.64 (3.41) | -2.01 (2.66)

5. Primary Outcome: Change in Circumference
Time Frame: baseline, 4 weeks
Population: Children and parents
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
cm
  Children Waist Circumference: number analyzed (Participants) | 14 | 14
  Children Waist Circumference | -1.53 (3.01) | -2.96 (4.04)
  Parents Waist Circumference: number analyzed (Participants) | 14 | 14
  Parents Waist Circumference | -1.94 (5.80) | -0.49 (5.73)
  Children Midarm Circumference: number analyzed (Participants) | 14 | 14
  Children Midarm Circumference | -2.02 (2.17) | -1.14 (1.63)
  Parents Midarm Circumference: number analyzed (Participants) | 14 | 14
  Parents Midarm Circumference | -1.32 (2.06) | 0.35 (3.16)

6. Primary Outcome: Change in PAQ (Physical Activity Questionnaire)
Description: PAQ self reported questions based on activity level from 1 (low activity) to 5 (high activity), overall PAQ score is a mean of the questions.
Time Frame: baseline, 4 weeks
Population: Children
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 14 | 14
units on a scale | 0.22 (0.53) | -0.16 (0.54)

7. Primary Outcome: Change in Lipid Profile
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
mg/dL
  total cholesterol children: number analyzed (Participants) | 14 | 14
  total cholesterol children | -22.50 (36.31) | -16.50 (28.19)
  triglycerides children: number analyzed (Participants) | 14 | 14
  triglycerides children | -25.50 (95.26) | -13.14 (36.19)
  high-density lipoprotein cholesterol children: number analyzed (Participants) | 14 | 14
  high-density lipoprotein cholesterol children | -5.93 (9.37) | -2.93 (3.71)
  low-density lipoprotein cholesterol children: number analyzed (Participants) | 14 | 14
  low-density lipoprotein cholesterol children | -13.14 (35.54) | -11.00 (23.31)
  total cholesterol parents: number analyzed (Participants) | 14 | 14
  total cholesterol parents | -33.79 (30.84) | -7.14 (24.93)
  triglycerides parents: number analyzed (Participants) | 14 | 14
  triglycerides parents | 6.21 (41.71) | 16.86 (36.86)
  high-density lipoprotein cholesterol parents: number analyzed (Participants) | 14 | 14
  high-density lipoprotein cholesterol parents | -8.14 (41.71) | 16.86 (36.86)
  low-density lipoprotein cholesterol parents: number analyzed (Participants) | 14 | 14
  low-density lipoprotein cholesterol parents | -27.00 (26.72) | -5.50 (20.89)

8. Primary Outcome: Change in Glucose
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
mg/dL
  Children: number analyzed (Participants) | 14 | 14
  Children | 0.93 (6.01) | -.64 (5.02)
  Parent: number analyzed (Participants) | 14 | 14
  Parent | 4.93 (24.65) | -5.43 (12.40)

9. Primary Outcome: Change in hsCRP (High-sensitivity C-reactive Protein)
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
mg/L
  Children: number analyzed (Participants) | 14 | 14
  Children | -2.09 (7.10) | 2.78 (8.76)
  Parent: number analyzed (Participants) | 14 | 14
  Parent | -0.24 (1.36) | 0.21 (1.90)

10. Primary Outcome: Change in Liver Enzymes
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
U/L
  alanine aminotransferase (ALT) children: number analyzed (Participants) | 14 | 14
  alanine aminotransferase (ALT) children | 0.79 (14.35) | -1.14 (3.46)
  aspartate aminotransferase (AST) children: number analyzed (Participants) | 14 | 14
  aspartate aminotransferase (AST) children | 2.79 (8.96) | 0.00 (4.69)
  alanine aminotransferase (ALT) parents: number analyzed (Participants) | 14 | 14
  alanine aminotransferase (ALT) parents | 0.86 (7.01) | 4.57 (9.69)
  aspartate aminotransferase (AST) parents: number analyzed (Participants) | 14 | 14
  aspartate aminotransferase (AST) parents | 0.14 (5.70) | 4.43 (6.73)

11. Primary Outcome: Change in IL-6 (Interleukin-6)
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
pg/ml
  Children: number analyzed (Participants) | 14 | 14
  Children | -0.17 (0.89) | -0.19 (3.14)
  Parent: number analyzed (Participants) | 14 | 14
  Parent | 0.16 (0.90) | -0.19 (0.85)

12. Primary Outcome: Change in MPO (Myeloperoxidase)
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
pmol/L
  Children: number analyzed (Participants) | 14 | 14
  Children | -75.34 (37.34) | -69.23 (72.92)
  Parent: number analyzed (Participants) | 14 | 14
  Parent | 16.91 (110.66) | 1.78 (45.93)

13. Primary Outcome: Change in HgbA1c (Hemoglobin A1c)
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
percentage
  Children: number analyzed (Participants) | 14 | 14
  Children | 0.17 (0.17) | 0.21 (0.12)
  Parent: number analyzed (Participants) | 14 | 14
  Parent | -0.16 (0.16) | 0.14 (0.49)

14. Primary Outcome: Change in Insulin
Time Frame: baseline, 4 weeks
Population: Children and Parents
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Number analyzed (Participants) | 28 | 28
uU/ml
  Children: number analyzed (Participants) | 14 | 14
  Children | -5.42 (5.68) | 3.16 (25.62)
  Parents: number analyzed (Participants) | 14 | 14
  Parents | -3.11 (8.56) | -3.15 (5.47)

15. Secondary Outcome: PB/AHA - Adjusted Mean Difference BMI
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: percentile
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
percentile
  Children Change in BMI: number analyzed (Participants) | 28
  Children Change in BMI | -1.17 [-2.2 to -0.14]
  Parents Change in BMI: number analyzed (Participants) | 28
  Parents Change in BMI | -0.69 [-1.47 to 0.09]

16. Secondary Outcome: PB/AHA - Adjusted Mean Difference BMI Z Score Children
Time Frame: Baseline, 4 weeks
Population: Children
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | PB/AHA
Number analyzed (Participants) | 28
Z score | -0.13 [-0.24 to -0.03]

17. Secondary Outcome: PB/AHA - Adjusted Mean BP
Time Frame: Baseline, 4 weeks
Population: Children and parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children adj mean ratio systolic BP: number analyzed (Participants) | 28
  Children adj mean ratio systolic BP | 1.87 [-4.41 to 8.15]
  Children adj mean ratio diastolic BP: number analyzed (Participants) | 28
  Children adj mean ratio diastolic BP | 1.01 [0.92 to 1.11]
  parents adj mean ratio systolic BP: number analyzed (Participants) | 28
  parents adj mean ratio systolic BP | 0.97 [0.89 to 1.05]
  parents adj mean ratio diastolic BP: number analyzed (Participants) | 28
  parents adj mean ratio diastolic BP | 1.03 [0.94 to 1.13]

18. Secondary Outcome: PB/AHA - Adjusted Mean Difference Weight
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
kg
  Children Weight: number analyzed (Participants) | 28
  Children Weight | -1.71 [-3.80 to 0.39]
  Parents Weight: number analyzed (Participants) | 28
  Parents Weight | -1.95 [-4.16 to 0.26]

19. Secondary Outcome: PB/AHA - Adjusted Mean Difference Circumference
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
cm
  children waist circumference: number analyzed (Participants) | 28
  children waist circumference | 1.32 [-1.66 to 4.30]
  parents waist circumference: number analyzed (Participants) | 28
  parents waist circumference | -1.14 [-5.75 to 3.48]
  children arm circumference: number analyzed (Participants) | 28
  children arm circumference | -1.25 [-2.61 to 0.11]
  parents arm circumference: number analyzed (Participants) | 28
  parents arm circumference | -1.68 [-3.80 to 0.44]

20. Secondary Outcome: PB/AHA - Adjusted Mean Difference PAQ Children
Description: as for outcome 6
Time Frame: Baseline, 4 weeks
Population: Children
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PB/AHA
Number analyzed (Participants) | 28
units on a scale | 0.39 [-0.02 to 0.8]

21. Secondary Outcome: PB/AHA - Adjusted Mean Lipid Profile
Time Frame: Baseline, 4 weeks
Population: Children and parents
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
mg/dL
  CHOL children: number analyzed (Participants) | 28
  CHOL children | -10.34 [-36.48 to 15.8]
  TRIG children: number analyzed (Participants) | 28
  TRIG children | 1.01 [0.77 to 1.32]
  HDL children: number analyzed (Participants) | 28
  HDL children | 0.17 [-5.07 to 5.4]
  LDL children: number analyzed (Participants) | 28
  LDL children | 0.95 [0.8 to 1.13]
  CHOL parents: number analyzed (Participants) | 28
  CHOL parents | -27.29 [-48.68 to -5.9]
  TRIG parents: number analyzed (Participants) | 28
  TRIG parents | 0.95 [0.76 to 1.19]
  HDL parents: number analyzed (Participants) | 28
  HDL parents | 0.94 [0.87 to 1.02]
  LDL parents: number analyzed (Participants) | 28
  LDL parents | -21.92 [-40.37 to -3.46]

22. Secondary Outcome: PB/AHA - Adjusted Mean Ratio Glucose
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children: number analyzed (Participants) | 28
  Children | 1.01 [0.96 to 1.05]
  Parents: number analyzed (Participants) | 28
  Parents | 1.06 [0.97 to 1.16]

23. Secondary Outcome: PB/AHA - Adjusted Mean Ratio hsCRP
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children: number analyzed (Participants) | 28
  Children | 0.46 [0.21 to 1]
  Parents: number analyzed (Participants) | 28
  Parents | 0.68 [0.44 to 1.07]

24. Secondary Outcome: PB/AHA - Adjusted Mean Ratio Liver Enzymes
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  ALT children: number analyzed (Participants) | 28
  ALT children | 1 [0.76 to 1.32]
  AST children: number analyzed (Participants) | 28
  AST children | 1.13 [0.92 to 1.4]
  ALT parents: number analyzed (Participants) | 28
  ALT parents | 0.85 [0.67 to 1.08]
  AST parents: number analyzed (Participants) | 28
  AST parents | 0.83 [0.68 to 1.03]

25. Secondary Outcome: PB/AHA - Adjusted Mean Ratio IL-6
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children: number analyzed (Participants) | 28
  Children | 0.26 [0.05 to 1.37]
  Parents: number analyzed (Participants) | 28
  Parents | 1.14 [0.83 to 1.57]

26. Secondary Outcome: PB/AHA - Adjusted Mean Ratio MPO
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children: number analyzed (Participants) | 28
  Children | 0.95 [0.79 to 1.13]
  Parents: number analyzed (Participants) | 28
  Parents | 0.93 [0.8 to 1.1]

27. Secondary Outcome: PB/AHA - Adjusted Mean Ratio HgbA1c
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children: number analyzed (Participants) | 28
  Children | 0.99 [0.97 to 1.01]
  Parents: number analyzed (Participants) | 28
  Parents | 0.96 [0.92 to 1]

28. Secondary Outcome: PB/AHA - Adjusted Mean Ratio Insulin
Time Frame: Baseline, 4 weeks
Population: Children and Parents
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | PB/AHA
Number analyzed (Participants) | 56
ratio
  Children: number analyzed (Participants) | 28
  Children | 0.7 [0.43 to 1.12]
  Parents: number analyzed (Participants) | 28
  Parents | 0.87 [0.67 to 1.13]

ADVERSE EVENTS:
Arm/Group | Reduced Fat Vegan Diet | American Heart Association Diet
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No